CLINICAL TRIAL: NCT06120335
Title: Development and Reliability and Validity Evaluation of a Scale for Cancer Patients' Willingness to Voluntarily Participate in Drug Clinical Trials
Brief Title: Development of a Scale for Cancer Patients' Willingness to Voluntarily Participate in Drug Clinical Trials
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2023-1029-01
Record Dates: First submitted 2023-11-02; First posted 2023-11-07 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Cancer
Keywords: drug clinical trials; cancer patients; willingness
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to develop a scale for cancer patients' willingness to voluntarily participate in drug clinical trials and evaluate its reliability and validity.

DETAILED DESCRIPTION:
Inclusion Criteria:

1. Age 18-80 years old (including boundary values).
2. Tumor patients with clear diagnosis.
3. Whether they finally sign the informed consent form of one drug clinical trial or not, and whether they are finally enrolled in one drug clinical trial or not, patients who have undergone the informed consent process of drug clinical trials conducted by clinicians can be enrolled in this study.
4. Volunteer to participate in this study and sign an informed consent form.

Exclusion Criteria:

1. Patients with unclear consciousness.
2. Patients who are unable to correctly understand and answer questions.
3. Vulnerable subjects include: students and subordinates of researchers, military personnel, prisoners, patients with incurable diseases, patients in critical situations, those admitted to welfare institutions, homeless individuals, minors, and those who are unable to provide informed consent.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years old (including boundary values).
2. Tumor patients with clear diagnosis.
3. Whether they finally sign the informed consent form of one drug clinical trial or not, and whether they are finally enrolled in one drug clinical trial or not, patients who have undergone the informed consent process of drug clinical trials conducted by clinicians can be enrolled in this study.
4. Volunteer to participate in this study and sign an informed consent form.

Exclusion Criteria:

1. Patients with unclear consciousness.
2. Patients who are unable to correctly understand and answer questions.
3. Vulnerable subjects include: students and subordinates of researchers, military personnel, prisoners, patients with incurable diseases, patients in critical situations, those admitted to welfare institutions, homeless individuals, minors, and those who are unable to provide informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult tumor patients treated at Sun Yat sen Memorial Hospital at Sun Yat sen University
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-11-09 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
A semi-structured interview | 3 months
  A semi-structured interview is conducted to investigate the willingness of cancer patients to participate in drug clinical trials and its influencing factors. The researcher will analyze the interview results and summarize several themes that reflect the willingness.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong, China